CLINICAL TRIAL: NCT03191227
Title: The Cork and Kerry Diabetes and Heart Disease Study (Phase II)
Brief Title: The Cork and Kerry Diabetes and Heart Disease Study (Phase II) Mitchelstown Cohort
Acronym: Mitchelstown
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Livinghealth Clinic Mitchelstown (Unknown)
Responsible Party: Principal Investigator, Catherine Phillips, Dr Catherine Phillips, Senior Research Fellow and Co-Principal Investigator, University College Cork
Other Study IDs: HRC/2007/13
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Diseases; Diabetes; Obesity; Hypertension; Dyslipidemia; Metabolic Syndrome; Diet Habit; Life Style; Physical Activity; Smoking
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Hypertension; Dyslipidemias; Metabolic Syndrome; Feeding Behavior; Motor Activity; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the Cork and Kerry Study Phase II (Mitchelstown cohort recruited 2010-11) is to provide an updated profile of glucose tolerance status, cardiovascular health and their related factors in an Irish adult general population sample and to compare the findings with those obtained during baseline assessment of Phase I of the Cork and Kerry study (1998) and the rescreen (2008).

DETAILED DESCRIPTION:
Additional objectives include determining the prevalence of proximal risk factors, such as hypertension, dyslipidaemia, body mass index (BMI) and insulin resistance as well as of more distal risk factors of diet, smoking, alcohol consumption and physical activity, and the association between cardiovascular health and its risk factors with general measures of well-being and mental health. The new cohort includes collection of qualitative and quantitative data in an effort not only to describe the current health status of the cohort and assess individual level determinants but also to provide the appropriate context to interpret the role of behavioural factors and social circumstances on health.

Recruitment was completed on a new cohort of 2047 men and women aged 50-69 years from patients attending a single large primary care centre, the Living Health Clinic in Mitchelstown, a town with a population of 43000 in county Cork. The Living Health clinic includes eight GPs, and the practice serves a catchment area of 20 000, with a mix of urban and rural residents. Participants were randomly selected from all registered attending patients in the 50-69-year age group.

ELIGIBILITY:
Inclusion Criteria:

All participants from the Livinghealth Clinic practice list in the 50-69 year age bracket

Exclusion Criteria:

Duplicates, deaths and ineligibles and those who did not complete the general health questionnaire and physical examination

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment was completed on a new cohort of 2047 men and women aged 50-69 years from patients attending a single large primary care centre, the Living Health Clinic in Mitchelstown, a town with a population of 43000 in county Cork. The Living Health clinic includes eight GPs, and the practice serves a catchment area of 20 000, with a mix of urban and rural residents. Participants were randomly selected from all registered attending patients in the 50-69-year age group (response rate: 67%).
Sampling Method: Non-Probability Sample
Enrollment: 2047 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease | At baseline
  The presence of cardiovascular disease (CVD) was obtained from the GHQ by asking study participants if they had been diagnosed with any one of the following seven conditions: Heart Attack (including coronary thrombosis or myocardial infarction), Heart Failure, Angina, Aortic Aneurysm, Hardening of the Arteries, Stroke, or any other Heart Trouble. Subjects who indicated a diagnosis of any one of these conditions were classified as having CVD.
Type 2 Diabetes | At baseline
  Type 2 diabetes was defined according to the American Heart Association guidelines of fasting plasma glucose (FPG) ≥ 7 mmol/L or doctor diagnosed diabetes.
Obesity | At baseline
  Anthropometric measurements were recorded with calibrated instruments according to a standardised protocol. Body weight was measured in kilograms without shoes; to the nearest 100g using a Tanita WB100MA® weighing scales (Tanita Corporation, IL, USA). Height was measured in centimetres to one decimal place using a Seca Leicester® height gauge (Seca, Birmingham, UK). BMI was calculated as weight (kg) /height (m)2. Individuals with a BMI ≥ 30kg/m2 were defined as obese.
Hypertension | At baseline
  Blood pressure was measured according to the European Society of Hypertension Guidelines using an Omron M7 Digital BP monitor on the right arm, after a 5-minute rest in the seated position. The average of the second and third measurements was used for analyses. Hypertension was defined as average systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg or being on hypertensive medication.
Metabolic syndrome | At baseline
  This is a composite measure classified using a range of MetS definitions (National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) 2001, 2004, American Diabetes Association, International Diabetes Federation) based on the following features: Waist circumference (WC), Fasting plasma glucose (FPG), High density lipoprotein cholesterol (HDL-C), Triglycerides (TG) and Blood pressure (BP).

SECONDARY OUTCOMES:
Depressive symptoms | At baseline
  Depressive symptoms were assessed using the 20-item Centre for Epidemiologic Studies Depression Scale (CES-D) questionnaire which was designed to evaluate the frequency and severity of depressive symptoms. History of depression was assessed using the following questions: "Have you ever had depression?" Subjects were then asked "If yes, when did it start? In the last year/ 1-5 years ago/ >5 years ago." Data regarding antidepressant medication use were collected. In addition to use of the aforementioned screening tool, subjects who indicated a diagnosis of depression or current anti-depressant medication use were classified as having a mental health disorder.
Anxiety | At baseline
  Anxiety was assessed using the Hospital Anxiety and Depression Scale (HADS), using only the anxiety subscale. History of anxiety was assessed using the following questions: "Have you ever had anxiety?" Subjects were then asked "If yes, when did it start? In the last year/ 1-5 years ago/ >5 years ago." Data regarding antidepressant medication use were collected. In addition to use of the aforementioned screening tool, subjects who indicated a diagnosis of depression or anxiety or current anti-depressant medication use were classified as having a mental health disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Perry, MD, PhD, Principal Investigator — University College Cork

IPD SHARING:
Plan to Share IPD: No
All collected source data are maintained and stored at the study research office, in the Department of Epidemiology and Public Health, University College Cork. Specific proposals for future collaboration would be welcomed. Further information can be found on the research centre website, http://www.hrbchdr.com/ or through email to patricia.kearney@ucc.ie.

REFERENCES:
- [Background] Kearney PM, Harrington JM, Mc Carthy VJ, Fitzgerald AP, Perry IJ. Cohort profile: The Cork and Kerry Diabetes and Heart Disease Study. Int J Epidemiol. 2013 Oct;42(5):1253-62. doi: 10.1093/ije/dys131. Epub 2012 Sep 14. No abstract available. PMID 22984148
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed/22984148 — Cohort profile